CLINICAL TRIAL: NCT01484028
Title: Clinical Validation of Etafilcon A With Print and PVP Contact Lenses for Dark Eyes and Light Eyes
Brief Title: Evaluation of the Performance of Two Contact Lenses Compared to a Marketed Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-005094
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Refractive Ametropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EALE/1DM (Other): etafilcon A with PVP for light eyes worn during the first period of 7-9 days then etafilcon A control lens worn during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A control lens (1DM); Device: etafilcon A with print and PVP for light eyes (EALE)
- 1DM/EALE (Other): etafilcon A control lens worn during the first period of 7-9 days then etafilcon A with PVP for light eyes worn during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A control lens (1DM); Device: etafilcon A with print and PVP for light eyes (EALE)
- EADE/1DM (Other): etafilcon A with PVP for dark eyes worn during the first period of 7-9 days then etafilcon A control lens worn during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A control lens (1DM); Device: etafilcon A with print and PVP for dark eyes (EADE)
- 1DM/EADE (Other): etafilcon A control lens worn during the first period of 7-9 days then etafilcon A with PVP for dark eyes worn during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
  Interventions: Device: etafilcon A control lens (1DM); Device: etafilcon A with print and PVP for dark eyes (EADE)

INTERVENTIONS:
Device: etafilcon A control lens (1DM) — A marketed daily disposable contact lens
  Other Names: 1-DAY ACUVUE MOIST Brand Contact Lenses
Device: etafilcon A with print and PVP for light eyes (EALE) — A daily disposable contact lens
  Arms: 1DM/EALE; EALE/1DM
Device: etafilcon A with print and PVP for dark eyes (EADE) — A daily disposable contact lens
  Arms: 1DM/EADE; EADE/1DM

SUMMARY:
This study will serve to evaluate and compare the performance of two new lenses to a marketed lens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, female adult, at least 18 years of age, and no more than 34 years of age
* The subjects must be female, light eye Caucasian, Non-Hispanic, habitual soft contact lens wearer (both eyes) with light or dark eyes
* Must have rated the Concept Statement positively (i.e., a rating of 4 or 5).
* Optimal vertexed spherical equivalent distance correction must be between -1.00 and -4.00 diopters (D)
* Any cylinder power must be: <=0.75D
* Visual acuity must be best correctable to 20/25 or better for each eye
* Must have normal eyes (no ocular medications or ocular infection of any type)
* Must read and sign the Statement of Informed Consent
* Must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear
* Systemic disease, autoimmune disease, or use of medication which might interfere with contact lens wear
* Clinically significant (grade 3 or worse) corneal edema, corneal neovascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear
* Any ocular infection
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear
* Any color deficiencies (colorblindness) - to the best of the subject's knowledge
* Pregnancy or lactation
* Diabetes
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV)
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.
* Subject presents with one dark iris color and one light iris color.
* Subject has heterochromia iridis (a difference in color between parts of one iris).
* The subject must not be an employee or family member of the clinical study site.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Advanced Optometry, Mission Viejo, California
  - James R Dugue, Optometrist, Mission Viejo, California
  - Advance Eye Care, Pismo Beach, California
  - Golden Vision, Sarasota, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - Eye Care Associates, Bloomington, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - Vision Care, East Lansing, Michigan
  - Spectrum Eye Care, Jamestown, New York
  - Sacco Eye Group, Vestal, New York
  - The Eye Care Group, Grants Pass, Oregon
  - Dr. David W Ferris and Associates, Warwick, Rhode Island
  - Wishnow Sugar Group, Katy, Texas
  - Isthmus Eye Care, Middleton, Wisconsin
  - Snowy Range Cision Center, Laramie, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 275 enrolled subjects, 267 subjects were randomized and received the study article in the study. Two subjects were discontinued between the first and second periods.
Groups:
- 1DM/EADE: etafilcon A control lens worn daily during the first period of 7-9 days then etafilcon A for dark eyes worn daily during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
- 1DM/EALE: etafilcon A control lens worn daily during the first period of 7-9 days then etafilcon A for light eyes worn daily during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
- EADE/1DM: etafilcon A for dark eyes worn daily during the first period of 7-9 days then etafilcon A control lens worn daily during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
- EALE/1DM: etafilcon A for light eyes worn daily during the first period of 7-9 days then etafilcon A control lens worn daily during the second period of 7-9 days, with a 1-3 days of wash-out time between the 2 periods.
Period: Period 1
Arm/Group | 1DM/EADE | 1DM/EALE | EADE/1DM | EALE/1DM
Started | 66 | 70 | 64 | 67
Completed | 66 | 67 | 64 | 66
Not Completed | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Non-Compliance to Protocol | 0 | 1 | 0 | 1
Not completed — Lens Discomfort | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | 1DM/EADE | 1DM/EALE | EADE/1DM | EALE/1DM
Started | 66 | 67 | 64 | 66
Completed | 66 | 67 | 64 | 66
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all randomized subjects who worn at least one pair of study lenses.
Groups:
- All Subjects: All randomized subjects who worn at least one pair of study lenses.
Arm/Group | All Subjects
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 267
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.94 (4.654)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Monocular Visual Acuity
Description: Monocular distance Snellen visual acuity (VA) scores were coverted to the algorithm of the minimal angle of resolution (LogMAR) scale based on the following formula: LogMAR = Log10 (VA/20) - a*VAR, where Log10 = base 10 logarithm, VA = the Snellen denominator score, a = LogMAR stepsize coefficient and VAR = letter gained or missing in addition to the Snellen denominator score.
Time Frame: Dispensing
Population: Analysis was conducted on all randomized subjects who wore at least one pair of study lenses.
Measure: Mean (Standard Deviation); unit: LogMAR score
Units Other Than Participants: eyes
Groups:
- EADE/EALE: etafilcon A with embedded print and PVP for dark/light eyes to correct myopia.
- 1-DM: A marketed daily disposable contact lens to correct myopia.
Arm/Group | EADE/EALE | 1-DM
Number analyzed (Participants) | 264 | 265
Number analyzed (eyes) | 528 | 530
LogMAR score | -0.044 (0.0618) | -0.060 (0.0589)
Statistical Analysis 1: Comparison: EADE/EALE vs 1-DM; The alternative hypothesis is the monocular distance Snellen VA (LogMAR scale) of etafilcon A with embedded print and PVP for dark/light eyes is non-inferior to that of etafilcon A control lenses; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.05 LogMAR was used; Mixed Models Analysis; Least-square mean difference = 0.011, 95% CI 2-sided [0.004 to 0.017], Standard Error of Mean 0.0034

2. Primary Outcome: Lens Fit Acceptance
Description: The overall lens fit was evaluated by the Investigators for each eye whether it was acceptable (yes/no).
Time Frame: Dispensing
Population: Analysis was conducted on all randomized subjects who wore at least one pair of study lenses.
Measure: Number (95% Confidence Interval); unit: % of Eyes
Units Other Than Participants: eyes
Groups:
- 1-DM: A marketed daily disposable contact lenses to correct myopia.
Arm/Group | EADE/EALE | 1-DM
Number analyzed (Participants) | 264 | 265
Number analyzed (eyes) | 528 | 530
% of Eyes | 100 [98.3 to 100] | 100 [98.3 to 100]

3. Primary Outcome: Corneal Staining of Grade 3 or 4
Description: Corneal staining was graded using a 5-point scale; 0=None(no staining), 1=Trace, 2=Mild, 3=Moderate, and 4=Severe. Only those eyes with corneal staining grade >= 3 were reported.
Time Frame: After 7-9 days of lens wear
Population: Analysis was conducted on all randomized subjects who wore at least one pair of study lenses.
Measure: Number (95% Confidence Interval); unit: % of Eyes
Units Other Than Participants: eyes
Groups:
- 1-DM: A marketed daily disposable contact lenses to correct myopia, two were discontinued between the first and second periods.
Arm/Group | EADE/EALE | 1-DM
Number analyzed (Participants) | 264 | 263
Number analyzed (eyes) | 528 | 526
% of Eyes | 0 [0 to 1.7] | 0 [0 to 1.7]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded when the subjects were exposed to the Investigational lenses.
Groups:
- Etafilcon A With PVP for Dark/Light Eyes: A daily disposable contact lens to correct myopia.
- Etafilcon A Control Lenses: A marketed daily disposable contact lens to correct myopia.
Arm/Group | Etafilcon A With PVP for Dark/Light Eyes | Etafilcon A Control Lenses
Serious Adverse Events (participants affected / at risk) | 0/267 | 0/267
Other Adverse Events (participants affected / at risk) | 0/267 | 0/267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No